CLINICAL TRIAL: NCT04927299
Title: Confirmatory Study of the Efficacy and Safety of the Combination of Losartan / Chlorthalidone vs Losartan / Hydrochlorothiazide in the Treatment of Patients With Essential Arterial Hypertension
Brief Title: Efficacy and Safety of Losartan/Chlorthalidone vs Losartan/Hydrochlorothiazide in Essential Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30601-III-20(1)
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Essential Arterial Hypertension
Keywords: Hypertension; Blood pressure; Diuretic; Losartan; Chlorthalidone
MeSH Terms: conditions — Hypertension | interventions — Losartan; Chlorthalidone; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Losartan + chlorthalidone (Experimental): Administered orally, one tablet a day, for 2 months.
  Interventions: Drug: Losartan/Chlorthalidone in fixed dose
- Group B: Losartan + hydrochlorothiazide (Active Comparator): Administered orally, one tablet a day, for 2 months.
  Interventions: Drug: Losartan + hydrochlorothiazide in fixed dose

INTERVENTIONS:
Drug: Losartan/Chlorthalidone in fixed dose — 1 tablet, once a day of 50 mg/12.5 or 100 mg/ 25 mg
  Other Names: LOS/CHLORTHA
  Arms: Group A: Losartan + chlorthalidone
Drug: Losartan + hydrochlorothiazide in fixed dose — 1 tablet, once a day of 50 mg/12.5 or 100 mg/ 25 mg
  Other Names: LOS/HYDROCHLO
  Arms: Group B: Losartan + hydrochlorothiazide

SUMMARY:
Phase IIIb, randomized, double-blind, prospective, multicenter study to evaluate the efficacy and safety of the fixed-dose combination of losartan / chlorthalidone compared with losartan / hydrochlorothiazide in the treatment of patients with essential arterial hypertension.

DETAILED DESCRIPTION:
Two groups of patients will be formed, who wil start treatment with the lower dose (Losartan 50 mg + chlorthalidone 12.5 mg; Losartan 50 mg + hydrochlorothiazide 12.5 mg).

Blood pressure (BP) figures will be evaluated and, in those patients who do not reach the therapeutic goal, defined as a decrease in Systolic blood pressure (SBP) / Diastolic blood pressure (DBP) values of 20/10 mmHg with respect to their baseline values or BP <140 / 90 mmHg, the dose will be escalated to the next available concentration for both treatments (Losartan 100 mg + chlorthalidone 25 mg; Losartan 100 mg + hydrochlorothiazide 25 mg) at 30 days or during an unscheduled visit.

After two months of treatment, the BP figures obtained with the final dose and the proportion of subjects who achieved a decrease in SBP / DBP values of 20/10 mmHg or <140/90 mmHg with respect to both combinations will be compared, and the frequency of adverse events presented will be described.

ELIGIBILITY:
Inclusion Criteria:

* Any sex.
* That they agree to participate in the study and give their informed consent in writing.
* Age between 18 and 65 years old at the beginning of the study.
* Patients with essential arterial hypertension with BP ≥140 / 90 mmHg and <180/110 mmHg.
* Women of childbearing potential using a contraceptive method (barrier, oral hormonal, injectable, subdermal), menopausal or surgically sterile.

Exclusion Criteria:

* The drug is contraindicated for medical reasons.
* Glomerular filtration rate ≤30 ml / min x 1.73 m2.
* Hypersensitivity to any of the components of the formula or other sulfonamides.
* Patients treated with other diuretics.
* Patient with a history of vascular disease (cerebrovascular disease, acute coronary syndrome, etc.) and acute renal failure in the last 6 months.
* Patient with severe complications of type 2 diabetes mellitus (Ketoacidosis or hyperosmolar nonketotic coma).
* Patients participating in another clinical study involving an investigational treatment or participated in one in the previous 4 weeks.
* Positive pregnancy test, women who are pregnant, breastfeeding or planning a pregnancy while conducting the study.
* Oncological patients (except basal cell skin cancer) or with serious diseases that, in the opinion of the investigator, have a serious prognosis or a life expectancy of less than 1 year, as well as mental illnesses.
* Patients diagnosed with gout.
* Patients whose participation in the study may be influenced (employment relationship with the research center or sponsor, inmates, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure (SBP) | Baseline and 2 months
  Evaluate the mean change in systolic blood pressure (SBP) at 2 months with respect to their baseline measurement, by treatment group with the final dose.
Change in diastolic blood pressure (DBP) | Baseline and 2 months
  Evaluate the mean change in diastolic blood pressure (DBP) at 2 months with respect to their baseline measurement, by treatment group with the final dose.

SECONDARY OUTCOMES:
Dosage adjustment requirement | 2 months
  Describe the proportion of subjects who required dose adjustment per treatment group.
Subjects who achieved blood pressure reduction goals | 2 months
  Proportion of subjects who decreased their systolic pressure by 20 mmHg and their diastolic pressure by 10 mmHg from baseline or blood pressure <140/90 mmHg per treatment group with the final dose.
Percentage of adherence to treatment | 2 months
  Assess the percentage of adherence to treatment during the intervention, by pill count.
Adverse events | 2 months
  Describe the frequency and intensity of adverse events and adverse reactions presented during the study by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J Zamora Muciño-Arroyo, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V. (BIOMED-AGS); Francisco Padilla Padilla, M.D, Principal Investigator — Independent; Juan A Peraza Zaldivar, M.D, Principal Investigator — Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V. (BIOMED-GDL); Luis M Román Pintos, PhD, Principal Investigator — Hospital Hispano S.A. de C.V.; Ernesto G Cardona Muñoz, M.D, Principal Investigator — Independent; Cinthia L Patiño Bernal, M.D, Principal Investigator — CICMEX Centro de Investigación Clínica de México S. de R.L. de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):e13-e115. doi: 10.1161/HYP.0000000000000065. Epub 2017 Nov 13. No abstract available. PMID 29133356
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Morales-Salinas A, Wyss F, Coca A, Ramirez AJ, Valdez O, Valerio LF. [Differences between the 2013 and 2014 hypertension guidelines.: Position of the Central American and Caribbean Society for Hypertension and Cardiovascular Prevention]. Rev Panam Salud Publica. 2015 Mar;37(3):172-8. Spanish. PMID 25988254
- [Background] 2018 ESC/ESH Guidelines for the management of arterial hypertension. Rev Esp Cardiol (Engl Ed). 2019 Feb;72(2):160. doi: 10.1016/j.rec.2018.12.004. No abstract available. English, Spanish. PMID 30704723
- [Background] Gonzalez-Juanatey JR, Mazon Ramos P. Cardiovascular prevention (VI). Use of drugs in the primary prevention of arterial hypertension and dyslipidemia. Rev Esp Cardiol. 2008 Aug;61(8):861-79. English, Spanish. PMID 18684369
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] Guerrero-Garcia C, Rubio-Guerra AF. Combination therapy in the treatment of hypertension. Drugs Context. 2018 Jun 6;7:212531. doi: 10.7573/dic.212531. eCollection 2018. PMID 29899755
- [Background] Ernst ME, Moser M. Use of diuretics in patients with hypertension. N Engl J Med. 2009 Nov 26;361(22):2153-64. doi: 10.1056/NEJMra0907219. No abstract available. PMID 19940300
- [Background] Kurtz TW, Klein U. Next generation multifunctional angiotensin receptor blockers. Hypertens Res. 2009 Oct;32(10):826-34. doi: 10.1038/hr.2009.135. Epub 2009 Aug 28. PMID 19713966
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Derived] Rucker-Joerg IE, Cardona-Munoz EG, Padilla-Padilla FG, Suarez-Otero R, Romero-Antonio Y, Canales-Vazquez E, Rios-Brito KF, Rodriguez-Vazquez IC, Gonzalez-Canudas J. Optimizing Blood Pressure Control: A Randomized Comparative Trial of Losartan/Chlorthalidone vs. Losartan/Hydrochlorothiazide. Cardiol Ther. 2025 Jun;14(2):231-247. doi: 10.1007/s40119-025-00407-7. Epub 2025 Apr 24. PMID 40274695
- See also: Official Journal of the Federation. PROJECT of Official Mexican Standard PROY-NOM-030-SSA2-2017, For the prevention, detection, diagnosis, treatment and control of systemic arterial hypertension. 2017. — http://www.dof.gob.mx/nota_detalle.php?codigo=5480159&fecha=19/04/2017
- See also: Official Mexican NORM NOM-008-SSA3-2017, For the comprehensive treatment of overweight and obesity. — http://www.dof.gob.mx/nota_detalle.php?codigo=5523105&fecha=18/05/2018